CLINICAL TRIAL: NCT00056563
Title: CSP #468 Phase I - A Comparison of Best Medical Therapy and Deep Brain Stimulation of Subthalamic Nucleus and Globus Pallidus for the Treatment of Parkinson's Disease
Brief Title: Phase I Deep Brain Stimulation (DBS) vs. Best Medical Therapy (BMT) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 468 Phase I; NCT00101556 (obsolete NCT alias)
Record Dates: First submitted 2003-03-18; First posted 2003-03-19 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; levo-dopa; tremor; dyskinesia; subthalamic nucleus; globus pallidus
MeSH Terms: conditions — Parkinson Disease; Tremor; Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Deep Brain Stimulation
  Interventions: Device: Bilateral Deep Brain Stimulation
- 2 (Active Comparator): Best Medical Therapy
  Interventions: Other: best medical therapy

INTERVENTIONS:
Device: Bilateral Deep Brain Stimulation — The DBS site (STN or GPi) will be assigned on a random basis at the time the patient enters the surgical phase of the trial.
  Arms: 1
Other: best medical therapy — Participants will initially be randomized to DBS or to 6 months of "best medical therapy." BMT participants will then proceed into the surgical phase of the trial. Effective 08/05/05, randomization to the BMT arm has been discontinued since the study has sufficient information to compare the outcomes of DBS and BMT patients at 6 months.
  Arms: 2

SUMMARY:
The goals of this study are to determine if simultaneous bilateral subthalamic nucleus stimulation or simultaneous bilateral globus pallidus stimulation is more effective in reducing symptoms of Parkinson's disease, and if deep brain stimulation or best medical therapy is more effective in improving Parkinson's disease symptoms

DETAILED DESCRIPTION:
Deep Brain Stimulation (DBS) is a promising therapy for Parkinson's disease (PD). Whether DBS is superior to comprehensive best medical therapy or whether some patients or symptoms respond better to DBS in one area of the brain or the other is currently not known. The goals of this project are to compare the effectiveness of DBS and comprehensive medical therapy as treatments for PD, and to compare bilateral DBS at 2 areas of the brain--the subthalamic nucleus (STN) and the globus pallidus (Gpi)--to determine the most effective brain site for surgical intervention In this prospective, randomized, multi-center trial, 316 patients will be enrolled at 13 centers over four and a half years. Patients will initially be randomized to immediate surgery (DBS) or to 6 months of "best medical therapy." BMT patients will then proceed into the surgical phase of the trial. The DBS site (STN or GPi) will be assigned on a random basis at the time the patient enters the surgical phase of the trial. Patients will be followed for two years post surgery (24-30 months). Effective 08/05/05, randomization to the BMT arm has been discontinued since the study has sufficient information to compare the outcomes of DBS and BMT patients at 6 months. The findings will be critically important in establishing the optimal surgical treatment of the disabling symptoms of PD.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson's disease,
* Hoehn and Yahr stage 2 or worse "off" medications,
* L-dopa responsive but with persistent disabling symptoms (i.e., refractory to "best medical treatment" with motor fluctuations, dyskinesias),
* on stable medical therapy for at least one month prior to enrollment,
* age > 21,
* available and willing to be followed-up according to study protocol, and
* no intracranial abnormalities that would contraindicate surgery (based on pre-operative magnetic resonance imaging of the brain).

Exclusion Criteria:

* "Parkinson's plus" syndromes,
* medical contraindications to surgery or stimulation,
* active alcohol or drug abuse,
* score on minimental status exam 24 or lower, or other neuropsychological dysfunction (e.g., dementia) that would contraindicate surgery,
* concurrent participation in another research protocol.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2002-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Follett, Study Chair — VA Medical Center, Iowa City; Frances M. Weaver, PhD MA BA, Study Chair — Edward Hines Jr. VA Hospital
Locations (14):
- United States (14):
  - University of California at Los Angeles, Los Angeles, California
  - VA Medical Center, San Francisco, San Francisco, California
  - University of California at San Francisco, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Medical Center, Iowa City, Iowa City, Iowa
  - VA Medical Center, Portland, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Medical College of Virginia, Richmond, Virginia
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

REFERENCES:
- [Result] Follett K, Weaver F, Stern M, Marks W, Hogarth P, Holloway K, Bronstein J, Duda J, Horn S, Lai E, Samii A. Multisite randomized trial of deep brain stimulation. Arch Neurol. 2005 Oct;62(10):1643-4; author reply 1644-5. doi: 10.1001/archneur.62.10.1643-b. No abstract available. PMID 16216957
- [Result] Weaver F, Follett K, Hur K, Ippolito D, Stern M. Deep brain stimulation in Parkinson disease: a metaanalysis of patient outcomes. J Neurosurg. 2005 Dec;103(6):956-67. doi: 10.3171/jns.2005.103.6.0956. PMID 16381181
- [Result] Weaver FM, Stern MB, Follett K. Deep-brain stimulation in Parkinson's disease. Lancet Neurol. 2006 Nov;5(11):900-1. doi: 10.1016/S1474-4422(06)70586-5. No abstract available. PMID 17052655
- [Result] Weaver FM, Follett K, Stern M, Hur K, Harris C, Marks WJ Jr, Rothlind J, Sagher O, Reda D, Moy CS, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein J, Stoner G, Heemskerk J, Huang GD; CSP 468 Study Group. Bilateral deep brain stimulation vs best medical therapy for patients with advanced Parkinson disease: a randomized controlled trial. JAMA. 2009 Jan 7;301(1):63-73. doi: 10.1001/jama.2008.929. PMID 19126811
- [Result] Genever RW. Deep brain stimulation for patients with advanced Parkinson disease. JAMA. 2009 May 20;301(19):1985; author reply 1985-6. doi: 10.1001/jama.2009.647. No abstract available. PMID 19454631
- [Result] Follett KA, Weaver FM, Stern M, Hur K, Harris CL, Luo P, Marks WJ Jr, Rothlind J, Sagher O, Moy C, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein JM, Stoner G, Starr PA, Simpson R, Baltuch G, De Salles A, Huang GD, Reda DJ; CSP 468 Study Group. Pallidal versus subthalamic deep-brain stimulation for Parkinson's disease. N Engl J Med. 2010 Jun 3;362(22):2077-91. doi: 10.1056/NEJMoa0907083. PMID 20519680
- [Result] Hou B, Jiang T, Liu R. Deep-brain stimulation for Parkinson's disease. N Engl J Med. 2010 Sep 2;363(10):987-8; author reply 988. doi: 10.1056/NEJMc1007650. No abstract available. PMID 20830819
- [Result] Bronstein JM, Tagliati M, Alterman RL, Lozano AM, Volkmann J, Stefani A, Horak FB, Okun MS, Foote KD, Krack P, Pahwa R, Henderson JM, Hariz MI, Bakay RA, Rezai A, Marks WJ Jr, Moro E, Vitek JL, Weaver FM, Gross RE, DeLong MR. Deep brain stimulation for Parkinson disease: an expert consensus and review of key issues. Arch Neurol. 2011 Feb;68(2):165. doi: 10.1001/archneurol.2010.260. Epub 2010 Oct 11. PMID 20937936
- [Derived] Ostrem JL, Luo P, Weaver FM, Follett K, Rothlind J, Galifianakis NB, Lai EC, Bronstein J, Duda J, Holloway K, Sarwar A, Brodsky M, Chung K, Spindler M, Reda D, Snodgrass A, Moy C, Huang G, Wei Y, Marks WJ Jr; CSP 468F Study Group. 10-year clinical outcomes of subthalamic nucleus versus pallidal deep brain stimulation for Parkinson's disease: VA/NINDS CSP #468F. Front Neurol. 2026 Jan 16;16:1728999. doi: 10.3389/fneur.2025.1728999. eCollection 2025. PMID 41626017
- [Derived] Rothlind JC, York MK, Carlson K, Luo P, Marks WJ Jr, Weaver FM, Stern M, Follett K, Reda D; CSP-468 Study Group. Neuropsychological changes following deep brain stimulation surgery for Parkinson's disease: comparisons of treatment at pallidal and subthalamic targets versus best medical therapy. J Neurol Neurosurg Psychiatry. 2015 Jun;86(6):622-9. doi: 10.1136/jnnp-2014-308119. Epub 2014 Sep 2. PMID 25185211
- [Derived] Weintraub D, Duda JE, Carlson K, Luo P, Sagher O, Stern M, Follett KA, Reda D, Weaver FM; CSP 468 Study Group. Suicide ideation and behaviours after STN and GPi DBS surgery for Parkinson's disease: results from a randomised, controlled trial. J Neurol Neurosurg Psychiatry. 2013 Oct;84(10):1113-8. doi: 10.1136/jnnp-2012-304396. Epub 2013 May 10. PMID 23667214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment begun in May 2002 and the discontinuation of randomization to the BMT arm was approved in August 2005 and participating sites received their IRB approval of this change through October 2005. A total of 255 patients were randomized to either BMT or DBS from 7 VA medical centers and 6 affiliated university sites.
Pre-assignment Details: An additional 23 patients were screened after signing the informed consent form but not randomized. 11 of them weren't willing to participate in the follow-up visits after intervention, 7 of them had neuropsychological dysfunction, 2 of them were not responsive to levodopa, and 3 had medical contraindication to surgery and/or DBS stimulation.
Groups:
- 1: Bilateral Deep Brain Stimulation: Bilateral Deep Brain Stimulation
  Bilateral Deep Brain Stimulation : The DBS site (STN or GPi) will be assigned on a random basis at the time the patient enters the surgical phase of the trial.
- 2: Best Medical Therapy: Best Medical Therapy
  best medical therapy : Participants will initially be randomized to DBS or to 6 months of
Period: Overall Study
Arm/Group | 1: Bilateral Deep Brain Stimulation | 2: Best Medical Therapy
Started | 121 | 134
Completed | 121 | 134
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2: Best Medical Therapy: Best Medical Therapy
  best medical therapy : Participants will initially be randomized to DBS or to 6 months of "best medical therapy." BMT participants will then proceed into the surgical phase of the trial. Effective 08/05/05, randomization to the BMT arm has been discontinued since the study has sufficient information to compare the outcomes of DBS and BMT patients at 6 months.
- Total: Total of all reporting groups
Arm/Group | 1: Bilateral Deep Brain Stimulation | 2: Best Medical Therapy | Total
Number analyzed (Participants) | 121 | 134 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 97 | 187
  >=65 years | 31 | 37 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (8.8) | 62.3 (9.0) | 62.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 98 | 110 | 208
Region of Enrollment [Number; unit: participants]
  United States | 121 | 134 | 255

OUTCOME MEASURES:

1. Primary Outcome: The Difference of Time Spent in the 'on' State Without Troublesome Dyskinesia Based on Patient Motor Diaries as Compared to the Baseline.
Time Frame: at six months
Measure: Mean (95% Confidence Interval); unit: Hours per day
Arm/Group | 1: Bilateral Deep Brain Stimulation | 2: Best Medical Therapy
Number analyzed (Participants) | 121 | 134
Hours per day | 4.6 [3.8 to 5.3] | 0 [-0.5 to 0.5]

2. Secondary Outcome: The Change of Scores on the UPDRS for Blinded Assessed Motor Function 'Off' Medication and 'on' Stimulation
Description: Unified Parkinson's Disease Rating Scale (UPDRS Part III) measured while the patient is off medications and on stimulation at follow-up visits post surgery. UPDRS Part III has 14 items assessing motor skills including facial expression and speech, tremors, rigidity, posture, gait, and bradykinesia. Left and right sides (arms, legs, and hands) are assessed separately for seven of the functions. A summary score ranging from 0 to 108 is generated by adding the 14 specific motor function responses. The motor function (UPDRS part III) assessments are done by turning on the stimulation with and without taking PD medications (on/off) at each in-person visit. The higher score indicates that the condition is worse.
Time Frame: at six months
Measure: Mean (95% Confidence Interval); unit: units
Arm/Group | 1: Bilateral Deep Brain Stimulation | 2: Best Medical Therapy
Number analyzed (Participants) | 121 | 134
units | -12.3 [-14.3 to -10.3] | -1.7 [-3.3 to -0.1]

ADVERSE EVENTS:
Arm/Group | 1: Bilateral Deep Brain Stimulation | 2: Best Medical Therapy
Serious Adverse Events (participants affected / at risk) | 49/121 | 15/134
Other Adverse Events (participants affected / at risk) | 116/121 | 97/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Bilateral Deep Brain Stimulation (N=121) | 2: Best Medical Therapy (N=134)
Surgical Site Infection (Surgical and medical procedures) | 12 (16) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Confusional State (Psychiatric disorders) | 3 (3) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Dyskinesia (Nervous system disorders) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (3) | 0 (0)
Procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Angina Unstable (Cardiac disorders) | 1 (1) | 1 (1)
Angioplasty, Bone Graft, transurethral prostatectomy (Surgical and medical procedures) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary disease, Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Deep Vein Thrombosis, Orthostatic hypertension (Vascular disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hallucination (Psychiatric disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Coronary Artery Insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Gastrooesopageal Reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Lethargy (General disorders) | 1 (1) | 0 (0)
Mechanical complication of implant (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Urinary Tract infection (Infections and infestations) | 1 (1) | 0 (0)
Complication of device removal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device migration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medical Device complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medical device discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Glioma, Lung Neoplasm malignant, Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Nervous system disorders (Nervous system disorders) | 15 (15) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Sexual Dysfunction (Psychiatric disorders) | 1 (1) | 0 (0)
Activities of daily living impaired (Social circumstances) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.7% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Bilateral Deep Brain Stimulation (N=121) | 2: Best Medical Therapy (N=134)
Fall (Injury, poisoning and procedural complications) | 49 (66) | 22 (25)
Motor Dysfunction (Nervous system disorders) | 26 (29) | 25 (25)
Dyskinesia (Nervous system disorders) | 37 (44) | 23 (23)
Tremor (Nervous system disorders) | 30 (37) | 22 (23)
Gait disturbance (Nervous system disorders) | 37 (41) | 21 (21)
Bradykinesia (Nervous system disorders) | 25 (29) | 20 (20)
Balance disorder (Nervous system disorders) | 22 (24) | 19 (19)
Dysphagia (Gastrointestinal disorders) | 32 (35) | 17 (19)
Muscle rigidity (Nervous system disorders) | 24 (27) | 17 (17)
Speech disorder (Nervous system disorders) | 34 (40) | 16 (16)
Orthostatic hypotension (Vascular disorders) | 27 (33) | 16 (17)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 23 (28) | 16 (18)
Confusional state (Psychiatric disorders) | 33 (41) | 15 (15)
Dystonia (Nervous system disorders) | 31 (37) | 15 (16)
Depression (Psychiatric disorders) | 28 (32) | 15 (16)
Pain (General disorders) | 27 (35) | 15 (15)
Freezing phenomenon (Nervous system disorders) | 31 (33) | 14 (14)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 18 (20) | 14 (14)
Akinesia (Nervous system disorders) | 14 (18) | 12 (13)
Headache (Nervous system disorders) | 40 (49) | 2 (2)
Constipation (Gastrointestinal disorders) | 23 (25) | 9 (9)
Incision site pain (General disorders) | 22 (23) | 0 (0)
Insomnia (Psychiatric disorders) | 20 (20) | 8 (8)
Procedural pain (Injury, poisoning and procedural complications) | 19 (22) | 0 (0)
Anxiety (Psychiatric disorders) | 16 (18) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 6 (6)
Drooling (Nervous system disorders) | 14 (14) | 6 (6)
Nausea (Gastrointestinal disorders) | 14 (15) | 3 (3)
Implant site infection (Infections and infestations) | 13 (18) | 0 (0)
Fatigue (General disorders) | 11 (12) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (2)

LIMITATIONS AND CAVEATS:
A limitation of this study is that the STN and GPi cases are pooled into a single DBS group. When the study was planned, it was thought that differences between STN and GPi at six months would be small, which was tested during the study analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other